CLINICAL TRIAL: NCT06921161
Title: Effectivity of TongueFit as Tongue Strength and Endurance Therapy in Children With Dysphagia: A Randomized Controlled Trial
Brief Title: Effectivity of TongueFit, A Novel Orofacial Manometer, as Tongue Strength and Endurance Therapy in Children With Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rizky Kusuma Wardhani (Other)
Responsible Party: Sponsor-Investigator, Rizky Kusuma Wardhani, Rizky Kusuma Wardhani, M.D., Physiatrist, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-02-0288
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dysphagia; Children
Keywords: dysphagia; effectivity; orofacial manometer; tongue strength; tongue endurance; children
MeSH Terms: conditions — Deglutition Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants (including parents of patients), physiatrists who conducted VFSS and physiatrists who examined the patients' tongue strength and endurance are all blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Oral Sensorimotor Stimulation Therapy
  Interventions: Other: OSMS
- Intervention group (Experimental): Combination Tongue Strength Exercise Therapy using TongueFit and OSMS Therapy
  Interventions: Device: TongueFit; Other: OSMS

INTERVENTIONS:
Device: TongueFit — TongueFit is a newly orofacial manometer. This device is specifically developed for children to measure and improve tongue strength and endurance which includes a complementary application. Participants will do a series of tongue exercise therapy using "TongueFit". The exercise therapy will be performed once per day, three times a week, for eight weeks.
  Other Names: Intervention; Orofacial manometer
  Arms: Intervention group
Other: OSMS — Patients will receive OSMS therapy, conducted for 15 minutes per session, three times a week, over a duration of eight weeks.
  Other Names: Control

SUMMARY:
The tongue plays a crucial role in the swallowing process, and weakness in its muscles can lead to difficulties in bolus control, mastication, bolus transport, and oral residue. Reduced tongue strength is closely associated with dysphagia, a swallowing disorder that impairs the movement of food or liquids from the mouth, pharynx, or esophagus into the stomach. Measuring tongue strength is essential not only for diagnosing dysphagia but also for setting therapeutic goals and evaluating treatment effectiveness.

However, Indonesia currently lacks accessible tools for assessing tongue strength and endurance or for providing tongue exercise therapy. Existing devices, such as the Tongueometer and Iowa Oral Performance Instrument (IOPI), are costly, difficult to access, and not well-suited for children. To address this gap, a prototype orofacial manometer (PMO) is needed-one that is affordable, child-friendly, and easy to use.

TongueFit is an innovative orofacial manometer designed for both assessing and improving tongue strength and endurance. Similar to the IOPI, this prototype provides objective measurements while also incorporating a biofeedback feature in the form of a video game, enhancing engagement and participation in therapy, particularly for children. Additionally, TongueFit offers advantages in affordability, accessibility, and usability. It has been validated as a reliable and accurate tool for measuring tongue function.

Given its potential, clinical trials are essential to evaluate the effectiveness of TongueFit in tongue strength and endurance therapy. These trials will support its broader clinical application and development, ensuring that it becomes a widely available tool for dysphagia management.

DETAILED DESCRIPTION:
This study was designed as a double-blinded and randomized controlled trial. Participants were selected through stratified random sampling. Upon meeting the inclusion and exclusion criteria, participants were randomly assigned to one of two groups (Intervention and Control Group). Each group consisted of 10 participants.

Participants in the control group received OSMS therapy, administered for 15 minutes per session, three times a week, over eight weeks. Participants in the intervention group received OSMS therapy combined with exercise therapy using the PMO "TongueFit." The exercise prescription followed the FITT principle (frequency, intensity, time, and type), incorporating both strengthening and endurance exercises. Strengthening exercises were performed at 60-80% intensity, while endurance exercises were performed at 40-60% intensity, with a frequency of 30 repetitions for each type. Each exercise session lasted 15 minutes and was conducted once per day, three times a week, for eight weeks.

Throughout the exercise therapy program, tongue strength and endurance measurements were taken every two weeks to adjust the target pressure needed for therapy. Evaluations for both groups were conducted at the 4th and 8th weeks, assessing tongue muscle strength and endurance. The mid- and final evaluation results were compared with baseline assessments to determine the effectiveness of each intervention method.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 16 years.
* Diagnosed with oral phase dysphagia based on VFSS, with an MBSImP score greater than 0 and ≤12.
* Ability to understand and follow instructions.
* Adequate postural control, demonstrated by the ability to maintain a sitting position and support the head.
* Good jaw stability (absence of open jaw posture, adequate lip seal).
* Parental consent and/or patient willingness to participate, confirmed through signed informed consent.

Exclusion Criteria:

* Children with multiple congenital craniomaxillofacial abnormalities.
* Children using visual aids (glasses) or hearing aids.
* Children with comorbid conditions that may deteriorate unpredictably.
* Patients currently receiving inpatient treatment.
* Children who are uncooperative during the training process.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Swallowing Function | Before enrollment of participants
  The examination was conducted using a Videofluoroscopic Swallowing Study (VFSS) to diagnose dysphagia by evaluating the Modified Barium Swallow Impairment Profile (MBSImP) score. The higher the score, the greater the disturbance.
Baseline Tongue Strength | At enrollment, the first meeting
  The force generated by the anteromedial elevation movement of the tongue creates contact between the anteromedial tongue and the hard palate and is measured in kilopascals (kPa).
Tongue Strength after 12 Sessions | 4th week (Middle of treatment)
  The force generated by the anteromedial elevation movement of the tongue creates contact between the anteromedial tongue and the hard palate and is measured in kilopascals (kPa).
Tongue Strength after 24 Sessions | 8th week (End of treatment)
  The force generated by the anteromedial elevation movement of the tongue creates contact between the anteromedial tongue and the hard palate and is measured in kilopascals (kPa).
Baseline Tongue Endurance | At enrollment, the first meeting
  The duration of the tongue ability to sustain submaximal pressure (50% of its maximum force)
Tongue Endurance after 12 sessions | 4th week (Middle of treatment)
  The duration of the tongue ability to sustain submaximal pressure (50% of its maximum force)
Tongue Endurance after 24 sessions | 8th week (End of treatment)
  The duration of the tongue ability to sustain submaximal pressure (50% of its maximum force)

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Medicine and Rehabilitation Polyclinic, Pediatric Division, Dr. Cipto Mangunkusumo Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No